CLINICAL TRIAL: NCT04620668
Title: Evaluating the Usefulness of an Artificial Intelligence (A.I.) Mental Health Chatbot in a Healthcare Setting
Brief Title: Can Mental Health Chatbots Help Chronic Disease Populations?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luke MacNeill (Other)
Collaborators: New Brunswick Innovation Foundation (Other); Touchkin eServices Pvt. Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Luke MacNeill, Postdoctoral Fellow, University of New Brunswick
Organization: University of New Brunswick (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: REB 036-2020
Record Dates: First submitted 2020-11-02; First posted 2020-11-09 (Actual); Results first posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-07

CONDITIONS: Arthritis; Diabetes; Depression; Anxiety; Stress
Keywords: Arthritis; Diabetes; Depression; Anxiety; Stress; Chatbot; Conversational Agent
MeSH Terms: conditions — Arthritis; Diabetes Mellitus; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of two groups. The treatment group will use a mental health chatbot (Wysa) over a period of four weeks. The control group will receive no intervention.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Wysa) (Experimental)
  Interventions: Device: Wysa
- Control Group (No Intervention)

INTERVENTIONS:
Device: Wysa — Wysa is an AI-based mental health chatbot. It uses evidence-based techniques to help users build mental resilience skills and improve their mental health.
  Arms: Treatment Group (Wysa)

SUMMARY:
Past research has shown that patients suffering from chronic health conditions tend to experience high levels of negative mental health symptoms (e.g., depression). The purpose of the current study is to evaluate whether an artificial intelligence (A.I.) mental health chatbot can be used to reduce negative mental health symptoms within this population. A minimum of 60 individuals with a chronic health condition (diabetes or arthritis) will be recruited. Participants will be randomly assigned to either a treatment group or a control group. Those assigned to the treatment group will use the mental health chatbot Wysa (Touchkin eServices, Bangalore) over a period of four weeks. Those assigned to the control group will receive no chatbot. Participants will complete measures of depression, anxiety, stress, and life satisfaction via Qualtrics at the outset of the study, two weeks into the study, and four weeks into the study (i.e., the final assessment point). Results from the treatment and control groups will be compared using ANOVA models. Participants in the treatment group will also be asked to complete some open-ended questions about their experiences with the chatbot program. A subset of participants from the treatment group may be asked to complete optional phone or video interviews to gain a better understanding of their experiences. Results will provide insight into the usefulness of chatbot programs for reducing negative mental health symptoms among patients with a chronic health condition. Results may also be used to inform policy decisions about the use of these programs for healthcare delivery, and to provide practical insight into how these programs can be best integrated into healthcare settings.

DETAILED DESCRIPTION:
People dealing with chronic health conditions are susceptible to mental health issues such as depression and anxiety. Providing conventional mental health services to all of these individuals is not practical given the limited resources of the healthcare system. Artificial intelligence (A.I.) mental health chatbots may be an accessible and cost-effective means by which people can receive some degree of mental health support while they cope with their conditions. These automated programs act as a source of virtual support, talking with individuals and providing them with therapeutic exercises to improve their mental wellbeing. Several chatbots have been designed to deliver interventions based on popular psychological therapies (e.g., Wysa, Woebot, and Tess). Research has shown that these programs can reduce symptoms of depression, anxiety, and stress in nonclinical populations. However, the effectiveness of these programs has not been tested in chronic disease populations.

The purpose of the current research is to gain a better understanding of the usefulness of mental health chatbots for chronic disease populations. This research will be guided by two fundamental objectives: (1) to determine whether a mental health chatbot can reduce or prevent negative mental health symptoms in individuals who are dealing with a chronic health condition, and (2) to learn more about how individuals with a chronic health condition view these programs, particularly in terms of their potential benefits or drawbacks when used in healthcare settings. This research will focus on two specific chronic disease populations that are prone to elevated levels of mental health symptoms: people with arthritis and diabetes.

Participants will be recruited through social media channels (including online groups), newspaper advertisements, and emails and newsletters from relevant organizations (e.g., the Arthritis Society, Diabetes Canada). After volunteering to participate, participants will set up a phone or video conferencing call with the primary investigator to orient them into the study. Participants will be randomly assigned to either a treatment group or control group. Those assigned to the treatment group will download the mental health chatbot Wysa (Touchkin eServices, Bangalore) on their smartphones. They will interact with the chatbot a minimum of two times per week over a period of four weeks, with each interaction lasting a minimum of five minutes. Participants assigned to the control group will receive no chatbot (i.e., they will be in a no-treatment control group).

Regardless of their group assignment, participants will complete online materials via Qualtrics at the outset of the study, two weeks into the study, and four weeks into the study (i.e., the final assessment point). At the outset of the study, participants will fill out an informed consent form, a demographic questionnaire, and four psychological assessments tools: measures of depression, anxiety, stress, and life satisfaction. Two weeks into the study, participants will complete the four psychological assessment tools a second time. Four weeks into the study, participants will complete the four assessment tools a final time, and those in the treatment group will be presented with a post-study questionnaire that contains qualitative questions regarding their experiences with the chatbot. Participants in both groups will be presented with a debriefing form providing more information about the study. Those in the control group will be given the opportunity to download and use the chatbot at this point.

After the data from the four-week study are analyzed, a subset of participants from the treatment group may be asked to complete optional phone or video interviews to gain more insight into their experiences with and opinions on the chatbot program. Approximately 15 to 20 participants will be sought for the interviews. The questions for these interviews will be developed based on the collective results from the quantitative and qualitative analysis described above.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a diagnosis of diabetes (type 1 or type 2 diabetes) or arthritis (osteoarthritis, rheumatoid arthritis, or another type of arthritis).
* Participants must have a phone with an active Internet connection.

Exclusion Criteria:

* Participants must not be receiving ongoing treatment from a mental health professional.
* Participants must not be using a mental health chatbot (i.e., prior to the study).
* Participants must not have started or experienced a dosage change in a psychopharmacological drug within the previous month.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luke MacNeill, PhD, Principal Investigator — Centre for Research in Integrated Care, University of New Brunswick
Locations (1):
- Centre for Research in Integrated Care, University of New Brunswick, Saint John, New Brunswick, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fitzpatrick KK, Darcy A, Vierhile M. Delivering Cognitive Behavior Therapy to Young Adults With Symptoms of Depression and Anxiety Using a Fully Automated Conversational Agent (Woebot): A Randomized Controlled Trial. JMIR Ment Health. 2017 Jun 6;4(2):e19. doi: 10.2196/mental.7785. PMID 28588005
- [Background] Fulmer R, Joerin A, Gentile B, Lakerink L, Rauws M. Using Psychological Artificial Intelligence (Tess) to Relieve Symptoms of Depression and Anxiety: Randomized Controlled Trial. JMIR Ment Health. 2018 Dec 13;5(4):e64. doi: 10.2196/mental.9782. PMID 30545815
- [Background] Inkster B, Sarda S, Subramanian V. An Empathy-Driven, Conversational Artificial Intelligence Agent (Wysa) for Digital Mental Well-Being: Real-World Data Evaluation Mixed-Methods Study. JMIR Mhealth Uhealth. 2018 Nov 23;6(11):e12106. doi: 10.2196/12106. PMID 30470676
- [Background] Ly KH, Ly AM, Andersson G. A fully automated conversational agent for promoting mental well-being: A pilot RCT using mixed methods. Internet Interv. 2017 Oct 10;10:39-46. doi: 10.1016/j.invent.2017.10.002. eCollection 2017 Dec. PMID 30135751
- [Background] Clarke DM, Currie KC. Depression, anxiety and their relationship with chronic diseases: a review of the epidemiology, risk and treatment evidence. Med J Aust. 2009 Apr 6;190(S7):S54-60. doi: 10.5694/j.1326-5377.2009.tb02471.x. PMID 19351294
- [Derived] MacNeill AL, Doucet S, Luke A. Effectiveness of a Mental Health Chatbot for People With Chronic Diseases: Randomized Controlled Trial. JMIR Form Res. 2024 May 30;8:e50025. doi: 10.2196/50025. PMID 38814681

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from October 2021 to October 2022.
Pre-assignment Details: 98 individuals were assessed for eligibility. 19 did not meet inclusion criteria. 79 were assigned to groups.
Groups:
- Control Group: No treatment control group.
Period: Overall Study
Arm/Group | Treatment Group (Wysa) | Control Group
Started | 41 | 38
Completed | 34 | 34
Not Completed | 7 | 4
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Ineligible despite claims at outset of the study | 1 | 0
Not completed — Removed before analysis: missing data | 2 | 0
Not completed — Removed before analysis: failed multiple quality check questions | 1 | 2
Not completed — Removed before analysis: statistical outlier | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group (Wysa) | Control Group | Total
Number analyzed (Participants) | 34 | 34 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.50 (11.00) | 42.24 (11.66) | 42.87 (11.27)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Men | 8 | 12 | 20
  Gender: Women | 26 | 21 | 47
  Gender: Transgender Men | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 25 | 25 | 50
  Race/Ethnicity: Black / African Canadian | 0 | 1 | 1
  Race/Ethnicity: Indigenous / First Nations | 1 | 2 | 3
  Race/Ethnicity: Hispanic / Latino | 1 | 0 | 1
  Race/Ethnicity: Asian / Pacific Islander | 5 | 4 | 9
  Race/Ethnicity: Middle Eastern | 0 | 0 | 0
  Race/Ethnicity: Other | 0 | 1 | 1
  Race/Ethnicity: Mixed Race or Ethnicity | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  Canada | 34 | 34 | 68
Chronic Diseases [Count of Participants; unit: Participants]
  Diabetes | 16 | 16 | 32
  Arthritis | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Changes in Depression as Measured by the Patient Health Questionnaire (PHQ-9)
Description: The Patient Health Questionnaire (PHQ-9) contains nine items, each of which is rated on a scale of 0 to 3. Ratings are summed for a composite score; the minimum score is 0 and the maximum score is 27. Higher scores indicate higher levels of depression.
Time Frame: Participants are assessed at baseline, two weeks into the study, and four weeks into the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group (Wysa) | Control Group
Number analyzed (Participants) | 34 | 34
units on a scale
  Baseline | 8.65 (6.03) | 7.82 (6.29)
  Week 2 | 7.18 (4.90) | 7.41 (5.88)
  Week 4 | 5.26 (4.11) | 7.56 (6.33)
Statistical Analysis 1: Comparison: Treatment Group (Wysa) vs Control Group; Test type: Superiority; p < 0.001, Mixed ANOVA; Assessing interaction between experimental group and time point
Statistical Analysis 2: Comparison: Treatment Group (Wysa); Test type: Superiority; p < 0.001, Repeated Measures ANOVA; Assessing change within treatment group (follow-up to Mixed ANOVA)
Statistical Analysis 3: Comparison: Treatment Group (Wysa); Test type: Superiority; p = 0.044, Dependent t-test (2-sided); Assessing change within treatment group from baseline to week 2 (follow-up to Repeated Measures ANOVA). Bonferroni-adjusted p value
Statistical Analysis 4: Comparison: Treatment Group (Wysa); Test type: Superiority; p = 0.001, Dependent t-test (2-sided); Assessing change within treatment group from week 2 to week 4 (follow-up to Repeated Measures ANOVA). Bonferroni-adjusted p value
Statistical Analysis 5: Comparison: Control Group; Test type: Superiority; p = 0.731, Repeated Measures ANOVA; Assessing change within control group (follow-up to Mixed ANOVA)

2. Primary Outcome: Changes in Anxiety as Measured by the Generalized Anxiety Disorder Scale (GAD-7)
Description: The Generalized Anxiety Disorder Scale (GAD-7) contains seven items, each of which is rated on a scale of 0 to 3. Ratings are summed for a composite score; the minimum score is 0 and the maximum score is 21. Higher scores indicate higher levels of anxiety.
Time Frame: Participants are assessed at baseline, two weeks into the study, and four weeks into the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group (Wysa) | Control Group
Number analyzed (Participants) | 34 | 34
units on a scale
  Baseline | 7.44 (5.37) | 6.09 (6.27)
  Week 2 | 5.85 (4.02) | 6.32 (6.66)
  Week 4 | 4.74 (3.30) | 6.56 (6.45)
Statistical Analysis 1: Comparison: Treatment Group (Wysa) vs Control Group; Test type: Superiority; p < 0.001, Mixed ANOVA; Assessing interaction between experimental group and time point
Statistical Analysis 2: Comparison: Treatment Group (Wysa); Test type: Superiority; p < 0.001, Repeated Measures ANOVA; Assessing change within treatment group (follow-up to Mixed ANOVA)
Statistical Analysis 3: Comparison: Treatment Group (Wysa); Test type: Superiority; p = 0.05, Dependent t-test (2-sided); [statistical method as in outcome 1, analysis 3]
Statistical Analysis 4: Comparison: Treatment Group (Wysa); Test type: Superiority; p = 0.024, Dependent t-test (2-sided); [statistical method as in outcome 1, analysis 4]
Statistical Analysis 5: Comparison: Control Group; Test type: Superiority; p = 0.674, Repeated Measures ANOVA; Assessing change within control group (follow-up to Mixed ANOVA)

3. Primary Outcome: Changes in Stress as Measured by the Perceived Stress Scale (PSS-10)
Description: The Perceived Stress Scale (PSS-10) contains ten items, each of which is rated on a scale of 0 to 4. Ratings are summed for a composite score; the minimum score is 0 and the maximum score is 40. Higher scores indicate higher levels of stress.
Time Frame: Participants are assessed at baseline, two weeks into the study, and four weeks into the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group (Wysa) | Control Group
Number analyzed (Participants) | 34 | 34
units on a scale
  Baseline | 19.00 (6.79) | 17.53 (8.83)
  Week 2 | 18.56 (6.57) | 17.47 (7.82)
  Week 4 | 17.06 (6.21) | 17.35 (7.93)
Statistical Analysis 1: Comparison: Treatment Group (Wysa) vs Control Group; Test type: Superiority; p = 0.159, Mixed ANOVA; Assessing interaction between experimental group and time point

4. Secondary Outcome: Changes in Life Satisfaction as Measured by the Satisfaction With Life Scale
Description: The Satisfaction with Life Scale contains five items, each of which is rated on a scale of 1 to 7. Scores are summed for a composite score; the minimum score is 5 and the maximum score is 35. Higher scores indicate higher levels of life satisfaction.
Time Frame: Participants are assessed at baseline, two weeks into the study, and four weeks into the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group (Wysa) | Control Group
Number analyzed (Participants) | 34 | 34
units on a scale
  Baseline | 18.91 (6.85) | 19.59 (7.06)
  Week 2 | 18.29 (6.87) | 19.50 (7.39)
  Week 4 | 20.29 (7.40) | 20.15 (6.94)
Statistical Analysis 1: Comparison: Treatment Group (Wysa) vs Control Group; Test type: Superiority; p = 0.326, Mixed ANOVA; Assessing interaction between experimental group and time point

ADVERSE EVENTS:
Time Frame: 4 weeks (from baseline assessment to final assessment)
Arm/Group | Treatment Group (Wysa) | Control Group
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/34
Serious Adverse Events (participants affected / at risk) | 1/34 | 1/34
Other Adverse Events (participants affected / at risk) | 1/34 | 2/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group (Wysa) (N=34) | Control Group (N=34)
Brief hospitalization (Surgical and medical procedures) | 1 | 0 — Brief hospitalization (unrelated to study).
Brief hospitalization (General disorders) | 0 | 1 — Brief hospitalization (unrelated to study).
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group (Wysa) (N=34) | Control Group (N=34)
Infectious disease (Infections and infestations) | 1 | 1 — Infectious disease (unrelated to study).
Dental procedure (Surgical and medical procedures) | 0 | 1 — Dental procedure (unrelated to study).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-13): https://cdn.clinicaltrials.gov/large-docs/68/NCT04620668/Prot_SAP_000.pdf